CLINICAL TRIAL: NCT01402128
Title: The Effect of Barley Beta-glucan on Serum Lipids and Body Weight
Brief Title: Efficacy and Safety of Fermented Barley on Decrement of Body Fat in Obese Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MTB-bG-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Results first posted 2012-12-25 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-11

CONDITIONS: Overweight; Hyperlipidemia
Keywords: Soluble fiber; Polycan; Overweight; LDL-C(Low Density Lipoprotein-cholesterol)
MeSH Terms: conditions — Overweight; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Barley beta-glucan(3.0g) (Experimental): Barley beta-glucan(3.0g/day) for 12 weeks
  Interventions: Dietary Supplement: Barley beta-glucan(3.0g)
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Barley beta-glucan(3.0g) — Barley beta-glucan(3.0g/day) for 12 weeks
  Arms: Barley beta-glucan(3.0g)
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
Barley, like oats, is a rich source of the soluble fibre β-glucan, which has been shown to significantly lower LDL-cholesterol (LDL-C). However, barley foods have been less widely studied.

DETAILED DESCRIPTION:
This study investigated whether the supplementation of barley β-glucan is reduce the visceral fat as well as the serum low-density lipoprotein cholesterol (LDL-C) and total cholesterol (TC) in mildly hypercholesterolemic subjects. In a 12 week double-blind, controlled study, subjects were randomized to one of treatment group(3.0g/day as β-glucan) or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* an age from 19 to 70 years,
* a BMI(Body Mass Index) >23 kg/m^2,
* an LDL-C(Low Density Lipoprotein-cholesterol) concentration between 110 and 250 mg/dL

Exclusion Criteria:

* they had heart disease, liver or kidney disease, food allergies, daily exercise habits, a body weight increase or decrease >10 kg in the previous 3 months, irregular lifestyle habits
* they took medication and functional foods known to affect lipid metabolism.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, MD., PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 19 to 70 years, BMI(Body Mass Index) >23 kg/m^2, and LDL-C(Low Density Lipoprotein-cholesterol) concentration between 110 and 250 mg/dL
Groups:
- Barley Beta-glucan: Barley beta-glucan(1times/day, 1packs/day, 3g/day) for 12weeks
  Barley beta-glucan: Barley as raw material is milled by crushing the liquefaction and saccharification enzymes reacted after baking yeast (S. cereviasiae) for 48 h, is produced through the fermentation process.
- Placebo: Placebo(1times/day, 1packs/day, 3g/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with Barley beta-glucan
Period: Overall Study
Arm/Group | Barley Beta-glucan | Placebo
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Barley Beta-glucan(3.0g) | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.7) | 48.5 (10.8) | 48.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Fat Mass(kg)
Description: Body fat mass(kg) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
kg
  Pre | 22.9 (4.4) | 24.3 (5.6)
  Post | 22.8 (4.8) | 24.1 (5.7)

2. Secondary Outcome: Changes in Visceral Adipose Tissue
Description: Visceral adipose tissue was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
cm^3
  Pre | 1250.7 (484.7) | 1296.1 (464.1)
  Post | 1140.3 (374.4) | 1165.7 (365.9)

3. Secondary Outcome: Changes in LDL-C (LDL Low Density Lipoprotein-cholesterol)
Description: LDL-C (LDL Low Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
mg/dl
  Pre | 141.7 (18.8) | 141.4 (28.5)
  Post | 141.7 (30.8) | 141.6 (31.4)

4. Secondary Outcome: Changes in HDL-C(High Density Lipoprotein-cholesterol)
Description: HDL-C(High Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
mg/dl
  Pre | 46.7 (9.7) | 47.1 (11.4)
  Post | 46.7 (12.3) | 46.1 (10.6)

5. Secondary Outcome: Changes in Total Cholesterol
Description: Total cholesterol was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
mg/dL
  Pre | 220.9 (23.5) | 220.0 (30.5)
  Post | 211.6 (35.2) | 210.9 (31.6)

6. Secondary Outcome: Changes in Triglyceride
Description: Triglyceride was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
mg/dL
  Pre | 141.9 (67.9) | 133.0 (55.7)
  Post | 141.1 (67.2) | 133.2 (62.7)

7. Secondary Outcome: Changes in FFA(Free Fatty Acid)
Description: FFA(free fatty acid) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: µEq/L
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
µEq/L
  Pre | 605.1 (243.8) | 591.1 (214.6)
  Post | 647.7 (194.3) | 644.4 (243.8)

8. Secondary Outcome: Changes in Apo-A1(Apolipoprotein A1)
Description: Apo-A1(Apolipoprotein A1) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
g/l
  Pre | 1.44 (0.20) | 1.42 (0.21)
  Post | 1.37 (0.25) | 1.36 (0.23)

9. Secondary Outcome: Changes in Apo-B(Apolipoprotein B)
Description: Apo-B(Apolipoprotein B) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
g/L
  Pre | 1.06 (0.16) | 1.05 (0.16)
  Post | 0.98 (0.19) | 0.99 (0.19)

10. Primary Outcome: Changes in Percent Body Fat(%)
Description: Percent body fat(%) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
percentage of body fat
  Pre | 33.1 (4.1) | 33.7 (4.6)
  Post | 33.1 (4.3) | 33.7 (4.7)

11. Secondary Outcome: Changes in Subcutaneous Adipose Tissue
Description: Subcutaneous adipose tissue was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Number analyzed (Participants) | 39 | 40
cm^3
  Pre | 2732.0 (603.4) | 2929.1 (792.6)
  Post | 2723.7 (644.7) | 2941.7 (817.3)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Barley Beta-glucan(3.0g) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No